CLINICAL TRIAL: NCT01948505
Title: Effect of IV Acetaminophen on Patients in the Neurocritical Care Unit
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00061838
Record Dates: First submitted 2013-09-18; First posted 2013-09-23 (Estimated); Results first posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2018-05

CONDITIONS: Post-operative Craniotomy Patients; Carotid Endarterectomy and Carotid Artery Stenosis Patients; Post-op Spine Patients Admitted to the NCCU; Endovascular Patients Undergoing Intracranial Intervention; Traumatic Brain Injuries NPO for at Least 12 Hours
Keywords: Craniotomy
MeSH Terms: interventions — Acetaminophen; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Active Comparator): IV acetaminophen: 1000mg IV q 8 hrs (scheduled) until: a) tolerating PO and IV saline-locked or b) 48 hours reached on medication
  Interventions: Drug: Intravenous acetaminophen
- Placebo Group (Placebo Comparator): IV Normal Saline: 100ml IV q 8 hrs (scheduled) until: a) tolerating PO and IV saline-locked or b) 48 hours reached on medication
  Interventions: Drug: Placebo for IV acetaminophen

INTERVENTIONS:
Drug: Intravenous acetaminophen
  Arms: Intervention group
Drug: Placebo for IV acetaminophen
  Other Names: Normal Saline
  Arms: Placebo Group

SUMMARY:
To assess the efficacy of an intravenous nonnarcotic pain medication on controlling patient pain.

To assess the effect of an intravenous nonnarcotic pain medication on patient sedation levels in neurocritically ill patients.

To assess the effect of an intravenous nonnarcotic pain medication on common side effects seen in patients taking other intravenous narcotic pain medication in the neurocritical care unit.

ELIGIBILITY:
Inclusion Criteria:

* > 45 kg (amenable to adult dosing)
* all traumatic brain injuries NPO for at least 12 hours
* all post-operative craniotomy patients
* all non-operative subarachnoid hemorrhage, intraparenchymal hemorrhage, and stroke patients
* all carotid endarterectomy and carotid artery stenosis patients
* all endovascular patients undergoing intracranial intervention
* all post-op spine patients admitted to the NCCU

Exclusion Criteria:

* documented allergy to acetaminophen
* documented severe hepatic impairment (Child-Pugh score > 6) or severe hepatic disease (hepatitis)
* documented severe renal impairment (CrCl < 30 ml/min) Blood tests will be performed prior to study procedures that will ensure patients do not have renal impairment.
* patients who are pregnant or breast feeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2013-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Sivakumar W, Jensen M, Martinez J, Tanana M, Duncan N, Hoesch R, Riva-Cambrin JK, Kilburg C, Ansari S, House PA. Intravenous acetaminophen for postoperative supratentorial craniotomy pain: a prospective, randomized, double-blinded, placebo-controlled trial. J Neurosurg. 2019 Mar 1;130(3):766-722. doi: 10.3171/2017.10.JNS171464. Epub 2018 Apr 20. PMID 29676689

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Group: IV acetaminophen: 1000mg IV q 8 hrs (scheduled) until: a) tolerating PO and IV saline-locked or b) 48 hours reached on medication
  Intravenous acetaminophen
- Placebo Group: IV Normal Saline: 100ml IV q 8 hrs (scheduled) until: a) tolerating PO and IV saline-locked or b) 48 hours reached on medication
  Placebo for IV acetaminophen
Period: Overall Study
Arm/Group | Experimental Group | Placebo Group
Started | 105 | 105
Completed | 105 | 105
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Placebo Group | Total
Number analyzed (Participants) | 102 | 102 | 204
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 50.6 [47.6 to 53.5] | 50.3 [47.4 to 53.2] | 50.5 [47.5 to 53.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 54 | 125
  Male | 31 | 48 | 79
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Narcotic Requirement After Surgery
Description: The primary efficacy end point was narcotic consumption during the first 48 hours after craniotomy. Opioid usage was calculated by converting the amount of the narcotics taken by the patient into oral morphine equivalents (ME), which were totaled for each postoperative day. At 48 hours after surgery, patients who received IV acetaminophen in addition to our standardized pain protocol did not have a statistically significantly lower mean narcotic requirement, measured in ME, when compared with those in the placebo group.
Time Frame: 48 hours
Measure: Mean (95% Confidence Interval); unit: Morphine Equivalents
Arm/Group | Experimental Group | Placebo Group
Number analyzed (Participants) | 102 | 102
Morphine Equivalents | 123.5 [102.9 to 144.2] | 134.2 [112.1 to 156.3]

2. Other Pre Specified Outcome: Frequency of Nausea, Vomiting, Urinary Retention & Constipation
Time Frame: 48 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Experimental Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/105
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/105
Other Adverse Events (participants affected / at risk) | 0/105 | 0/105

LIMITATIONS AND CAVEATS:
Caveats, a maximum of 3 g of IV acetaminophen was used to minimize the chance for acetaminophen-related toxicity and comply with current dosage recommendations of our university pharmacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No